CLINICAL TRIAL: NCT04531033
Title: Does Daily Supplementation of Lactobacillus Acidophilus MPH734 (Lacto-FreedomTM, or LF), for One Week, Affects Acute (Immediate), Subacute (7 Days), and Post-treatment Discontinuation (30-, 60-, and 90- Day) Lactose Metabolism, Gastrointestinal Symptoms, and Clinical Markers of Inflammation and Safety Compared to a Placebo?
Brief Title: Does Daily Supplementation of Lactobacillus Acidophilus MPH734, for One Week, Affect Acute (Immediate), Subacute (7 Days), and Post-treatment Discontinuation Lactose Metabolism, Gastrointestinal Symptoms, and Clinical Markers of Inflammation and Safety Compared to a Placebo
Acronym: LF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lemuel W. Taylor IV (Other)
Collaborators: Manzo Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Lemuel W. Taylor IV, Principal Investigator, University of Mary Hardin-Baylor
Organization: University of Mary Hardin-Baylor (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LF-1
Record Dates: First submitted 2020-08-18; First posted 2020-08-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lactose Intolerance
Keywords: lactose intolerance; probiotic
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Intervention Model Description: 3 treatments: low dose probiotic, high dose probiotic, placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Taken once prior to the first testing session, 3x a day every day for the 7 days of supplementation, and taken one last time during second testing session.
  Interventions: Dietary Supplement: Placebo
- Low dose 10 billion CFU per day (Experimental): Taken once prior to the first testing session, 3x a day every day for the 7 days of supplementation, and taken one last time during second testing session.
  Interventions: Dietary Supplement: Lactobacillus acidophilus MPH734
- High dose 15 billion CFU per day (Experimental): Taken once prior to the first testing session, 3x a day every day for the 7 days of supplementation, and taken one last time during second testing session.
  Interventions: Dietary Supplement: Lactobacillus acidophilus MPH734

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus MPH734 — After supplementing with oral probiotics, it has been suggested that select probiotics capable of expressing Beta-glucosidase enzyme activity may likewise be effective treatment for lactose intolerance.
  Other Names: Lacto-FreedomTM, or LF
  Arms: High dose 15 billion CFU per day; Low dose 10 billion CFU per day
Dietary Supplement: Placebo — placebo made to match dietary supplement being tested.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if twice or three times daily supplementation of Lactobacillus acidophilus MPH734 (Lacto-FreedomTM, or LF), for one week, affects acute (immediate), subacute (7 days), and post-treatment discontinuation (30-, 60-, and 90- day) lactose metabolism, gastrointestinal symptoms, and clinical markers of inflammation and safety compared to a placebo.

DETAILED DESCRIPTION:
Participants will be included and/or excluded in the study based on the criteria below:

Inclusion Criteria

* Participants will be male or female between the ages of 18-55 years;
* Participants will be apparently healthy and free from disease, as determined by a health history questionnaire;
* Participants will not be excluded if he or she has been clinically diagnosed with a carbohydrate malabsorption disorder, or is or has been prescribed to take prescription or over-the-counter medication for such;
* Participant has self-diagnosed or otherwise avoids consuming dairy, lactose, and other dairy-containing products, or regularly consumes Lactase enzymes for digestive support;
* Participant agrees and can comply with the study protocol;
* Participant provides signed and dated informed consent to participate in the study.

Subject Exclusion Criteria

* Participant is or may be pregnant, is trying to become pregnant, or is breastfeeding;
* Participant is insulin-dependent or -independent diabetic.
* Participant currently uses, or has discontinued the use of nicotine-containing products within twelve (12) months of the start of the study;
* Participant lives or works within an environment that chronically exposes the subject to second-hand smoke;
* Participant currently uses, or has discontinued the use of recreational drugs or medicinal marijuana within twelve (12) months of the start of the study;
* Participant has been clinically diagnosed with a digestive disorder such as gastrointestinal disease, chronic diarrhea or constipation, irritable or inflammatory bowel syndrome, Crohn's disease, or is, or has been prescribed to take prescription or over-the-counter medication for such;
* Participant has ever undergone gastric bypass surgery, or has undergone an abdominal or other gastrointestinal surgery within twelve (12) months of the start of the study;
* Participant is taking, or has taken antibiotic medications within two (2) weeks of the start of the study;
* Participant has undergone a colonoscopy within two (2) weeks of the start of the study, or is scheduled to receive a colonoscopy during the study;
* Participant has undergone a barium study or received an enema within two (2) weeks of the start of the study, or is scheduled to, or receives such during the study;
* Participant is taking, or has taken probiotics within two (2) weeks of the start of the study;
* Participant uses lactose digesting enzymes during the study;
* Participant is taking, or has taken weight loss, prebiotic [e.g., fructo- or galacto-oligosaccharides (FOS or GOS), psyllium, or insulin fiber, etc.], or laxative / stool softener dietary supplements, over-the-counter, or prescription medications within two (2) weeks of the start of the study;
* Participant is allergic to any ingredient present within the dietary supplement or placebo treatment;
* Participant reports any unusual adverse events associated with this study that, in consultation with the study investigators or the participant's doctor recommends removal from the body;
* Participant fails to comply with the study protocol.

Intervention Below is an overview of the study, including the phases, timepoints, and dependent variables that will be assessed. The total study duration for each subject is approximately fifteen (15) weeks - one (1) week of pre-test familiarization plus fourteen (14) weeks of intervention and testing. Subject testing will commence on a rolling enrollment basis (i.e., all subjects will not start, be tested on, and end the study at the same time).

24 hrs - 12 hrs: Restricted Diet

Discontinue eating:

* All grains (including pasta, bread, cereals)
* Fruits
* Vegetables (including any food products that contain corn, corn starch, etc)
* Nuts and seeds
* Beans/ Legumes
* All dairy products (including cheese, ice cream, butter, and yogurt)
* All meats [except those approved (below)]

Allowed foods:

* Baked or broiled chicken, fish or turkey (salt and pepper seasoning only)
* Plain, steamed white rice
* Eggs
* Clear chicken or beef broth
* White bread (only)
* Participants may drink water, coffee, or tea; no sugar or artificial sweetener; no creamer/cream 12 hrs - 0 hrs: Fasting
* Water only
* No sleeping or vigorous exercise for at least (1) hour prior to any time during the breath test

TIMELINE:

Day -7 - 0 - Pre-screening & Familiarization

* Subjects complete one-week nutrition log via MyFitnessPal Day 0 - Baseline & Acute Response (Lab Test #1; LT1)
* Subject arrives 12-hr fasted (water only) and having followed the 24hr pre-test and lifestyle protocol -> Body Mass (BM) and Hydration (urine) measurements -> 5-minute seated -> Heartrate (HR) and Blood Pressure (BP) measurements -> Gastrointestinal Symptom Score -> Venous Blood collection -> Non-Alcohol Mouth Rinse -> Breath Analysis -> Treatment Dose Consumed with 8-10 fl. oz. H2O -> 30- minute seated -> 25-gram Lactose Challenge/Ingestion -> 60- minute seated -> Non-Alcohol Mouth Rinse -> Breath Analysis -> 60-minute seated -> Non-Alcohol Mouth Rinse -> Breath Analysis -> 60 minute seated -> Gastrointestinal Symptoms Score -> Non-Alcohol Mouth Rinse -> Breath Analysis Day 1 - Day 7 - Treatment Phase
* Subjects consume three (3) servings per day of treatment at scheduled times and conditions for three (3) days -> On Day 4 subjects perform a Lactose Challenge / Ingestion Test at home after a12-hr fast (water only); Gastrointestinal Symptoms Score is collected prior to, and at 180 minutes postprandial (after lactose ingestion) -> Subjects continue to consume three (3) servings per day of treatment at scheduled times and conditions for three (3) days
* Subjects complete one-week nutrition log Day 7 - Subacute Response (Lab Test #2; LT2)
* Repeat LT1
* Subjects discontinue treatment Day 8 - Day 37 - 30- Day Post Treatment Phase
* Subjects perform weekly Lactose Challenge/Ingestion Testing at home with Gastrointestinal Symptoms Scoring
* Subjects complete one-week nutrition logs Day 37 - 30-Day Post Treatment Response (Lab Test #3; LT3)
* Repeat LT1/LT2 testing (less the Treatment Dose + 30-minute seating pre-Lactose Challenge / Ingestion) Day 38 - Day 67 - 60-Day Post Treatment Phase
* Subjects perform weekly Lactose Challenge/Ingestion Testing at home with Gastrointestinal Symptoms scoring
* Subjects complete one-week nutrition logs Day 67 - 60- Day Post Treatment Response (Lab Test #4; LT4)
* Repeat LT1/LT2/LT3 testing (less treatment Dose + 30-minute seated pre- Lactose Challenge/Ingestion) Day 68 - Day 97 - 90-Day Treatment Phase
* Subjects perform weekly Lactose Challenge/Ingestion Testing at home with Gastrointestinal Symptoms Scoring
* Subjects complete one-week nutrition logs Day 97 - 90-Day Post Treatment Response (Lab Test #5; LT5)
* Repeat LT1/LT2/LT3/LT4/ testing (less Treatment Dose + 30- minute seating pre- Lactose Challenge/ Ingestion)

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male or female between the ages of 18-55 years;
* Participants will be apparently healthy and free from disease, as determined by a health history questionnaire;
* Participants will not be excluded if he or she has been clinically diagnosed with a carbohydrate malabsorption disorder, or is or has been prescribed to take prescription or over-the-counter medication for such;
* Participant has self-diagnosed or otherwise avoids consuming dairy, lactose, and other dairy-containing products, or regularly consumes Lactase enzymes for digestive support;
* Participant agrees and can comply with the study protocol;
* Participant provides signed and dated informed consent to participate in the study.

Exclusion Criteria:

* Participant is or may be pregnant, is trying to become pregnant, or is breastfeeding;
* Participant currently uses, or has discontinued the use of nicotine-containing products within twelve (12) months of the start of the study;
* Participant lives or works within an environment that chronically exposes the subject to second-hand smoke;
* Participant currently uses, or has discontinued the use of recreational drugs or medicinal marijuana within twelve (12) months of the start of the study;
* Participant has been clinically diagnosed with a digestive disorder such as gastrointestinal disease, chronic diarrhea or constipation, irritable or inflammatory bowel syndrome, Crohn's disease, or is, or has been prescribed to take prescription or over-the-counter medication for such;
* Participant has ever undergone gastric bypass surgery, or has undergone an abdominal or other gastrointestinal surgery within twelve (12) months of the start of the study;
* Participant is taking, or has taken antibiotic medications within two (2) weeks of the start of the study;
* Participant has undergone a colonoscopy within two (2) weeks of the start of the study, or is scheduled to receive a colonoscopy during the study;
* Participant has undergone a barium study or received an enema within two (2) weeks of the start of the study, or is scheduled to, or receives such during the study;
* Participant is taking, or has taken probiotics within two (2) weeks of the start of the study;
* Participant uses lactose digesting enzymes during the study;
* Participant is taking, or has taken weight loss, prebiotic [e.g., fructo- or galacto-oligosaccharides (FOS or GOS), psyllium, or insulin fiber, etc.], or laxative / stool softener dietary supplements, over-the-counter, or prescription medications within two (2) weeks of the start of the study;
* Participant is allergic to any ingredient present within the dietary supplement or placebo treatment;
* Participant reports any unusual adverse events associated with this study that, in consultation with the study investigators or the participant's doctor recommends removal from the study;
* Participant fails to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Lactobacillus Acidophilus MPH734's Effect on lactose digestion in individuals who identify as lactose sensitive, intolerant, or avoid dairy. | 97 days
  Primary outcome of this study is to determine if twice or three times daily supplementation of Lactobacillus acidophilus MPH734 (Lacto-FreedomTM, or LF), for one week, affects acute (immediate), subacute (7 days), and post-treatment discontinuation (30-, 60-, and 90- day) lactose metabolism, gastrointestinal symptoms, and clinical markers of inflammation and safety compared to a placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mary Hardin-Baylor, Belton, Texas, United States